CLINICAL TRIAL: NCT00001981
Title: Acromegaly Treatment and Natural History
Brief Title: The Treatment and Natural History of Acromegaly
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 850082; 85-DK-0082
Record Dates: First submitted 2000-01-21; First posted 2000-01-24 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Acromegaly; Pituitary Neoplasm
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with acromegaly: Patients with acromegaly

SUMMARY:
The purpose of this study is to investigate the treatment and natural history of acromegaly. We have a longstanding interest in acromegaly treatment, and a cohort that has been followed for 30 years, or more in some cases. We will continue to follow patients and recruit new patients for treatment and follow-up. Blood and pituitary tumor tissue (when available through clinical care) will be saved for future analyses related to acromegaly.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the treatment and natural history of acromegaly. We have a longstanding interest in acromegaly treatment, and a cohort that has been followed for 30 years, or more in some cases. We will continue to follow patients and recruit new patients for treatment and follow-up.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be enrolled who are 18 years of age or over who are referred for care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involved patients who were referred to us and had acromegaly.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 1991-10-02 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
resolution of IGF-1 Growth Hormone abnormality | every 6 months & at end of study
  resolution of IGF-1 abnormality

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Gorden, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1985-DK-0082.html